CLINICAL TRIAL: NCT02761317
Title: Optimal Bowel Preparation Regimen for Patients With With a History of Colorectal Resection Before Colonoscopy
Brief Title: Optimal Bowel Preparation Regimen in Patients With Colorectal Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, PhD, MD, Shandong University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016SDU-QILU-03
Record Dates: First submitted 2016-04-28; First posted 2016-05-04 (Estimated); Last update posted 2016-06-02 (Estimated); Status verified 2016-05

CONDITIONS: Bowel Preparation
Keywords: bowel preparation; bisacodyl; polyethyleneglycol; colorectal surgery
MeSH Terms: interventions — Reference Standards; Bisacodyl

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- GroupA：standard preparation (Active Comparator): Subjects who are randomized into group A receive standard bowel preparation (2L PEG-ELS) on the same-day of procedure.
  Interventions: Drug: standard preparation (2L PEG-ELS)
- Group B:low-volume preparation (Experimental): Subjects who are randomized into group B receive 10mg bisacodyl at 6 pm on the evening before the colonoscopy and 2L PEG-ELS on the same-day of procedure. ( 2L PEG-ELS and 10mg bisacodyl )
  Interventions: Drug: low-volume preparation (10 mg bisacodyl plus 2L PEG-ELS)
- Group C：high-volume preparation (Experimental): Subjects who are randomized into group C will receive 2L PEG-ELS at 6 pm before the procedure and another 2L PEG-ELS on the same-day of procedure. (4 L PEG-ELS)
  Interventions: Drug: high-volume preparation (4L PEG-ELS)

INTERVENTIONS:
Drug: standard preparation (2L PEG-ELS) — Subjects who are randomized into group A will receive standard bowel preparation (2L PEG-ELS) on the same-day of procedure.
  Arms: GroupA：standard preparation
Drug: low-volume preparation (10 mg bisacodyl plus 2L PEG-ELS) — Subjects who are randomized into group B will receive 10mg bisacodyl at 6 pm on the evening before the colonoscopy and 2L PEG-ELS on the same-day of procedure.
  Arms: Group B:low-volume preparation
Drug: high-volume preparation (4L PEG-ELS) — Subjects who are randomized into group C will receive 2L PEG at 6 pm before the procedure and another 2L PEG-ELS on the same-day of procedure.(4L PEG)
  Arms: Group C：high-volume preparation

SUMMARY:
The study compares the efficacy of bowel cleansing between the standard preparation (2 L polyethylene glycol electrolyte solution, 2 L PEG-ELS), low-volume preparation (10 mg bisacodyl plus 2 L PEG-ELS) and high-volume preparation (4 L PEG-ELS) in patients with previous colorectal resection.

DETAILED DESCRIPTION:
Colonoscopy is the standard approach for evaluating the colon currently. Thorough bowel cleansing is critical for adequate visualization of colonic mucosa during colonoscopy. Inadequate bowel cleansing results in adverse consequences for the examination, including lower adenoma detection rates, longer procedural time, lower cecal intubation rates, shorter intervals between examinations and an estimated 12-22% increase in overall colonoscopy cost. A history of colorectal resection represents an independent predictor for inadequate colon cleansing,hence strategies to improve bowel preparation may be a demanding goal in this subset of patients.

The study compares the efficacy of bowel cleansing between the standard preparation (2 L polyethylene glycol electrolyte solution, 2 L PEG-ELS), low-volume preparation (10 mg bisacodyl plus 2 L polyethylene glycol electrolyte solution) and high-volume preparation (4L polyethylene glycol electrolyte solution, 4L PEG-ELS) in patients with previous colorectal resection. Then the investigators can select the optimized regimen for patients with colorectal surgery.

ELIGIBILITY:
Inclusion Criteria:

* All adults (18< age<75years) referred for surveillance colonoscopy with a history of colorectal resection for Colorectal cancer (CRC).

Exclusion Criteria:

* severe comorbidities (e.g. congestive heart failure and severe kidney disease)
* abdominal and pelvic surgery other than colorectal resection for the cause of CRC.
* severe colonic stricture or obstructing tumour
* dysphagia
* compromised swallowing reflex or mental status
* significant gastroparesis or gastric outlet obstruction
* known or suspected bowel obstruction or perforation
* severe chronic renal failure (creatinine clearance<30 ml/min
* severe congestive heart failure (New York Heart Association class III or IV)
* uncontrolled hypertension (systolic blood pressure>170 mm Hg, diastolic blood pressure>100 mm Hg)
* inflammatory bowel disease or megacolon
* dehydration
* disturbance of electrolytes
* pregnancy or lactation
* haemodynamically unstable
* unable to give informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2016-05; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Difference of scores rating by Aronchick Preparation Scale among 3 groups. | 6 months
  This is an established rating scale to evaluate the quality of bowel prep. The ratings will be compared among the 3 groups.

SECONDARY OUTCOMES:
Rate of compliance with instructions among 3 groups | 6 months
  Compliance was scored on a 3-grade scale based on the intake of bowel solution: 0 = optimal (intake of 100% of the solution); 1 = good (intake of ≥75% of the solution); 2 = poor (intake of <75% of the solution).
Willingness to repeat bowel preparation among 3 groups. | 6 months
  the willingness to repeat the same bowel preparation,a patient's subjective evaluation of the bowel preparation was recorded by a questionnaire
Polyp detection rate among 3 groups. | 6 months
  Polyp detection rate was defined as the proportion of patients with at least one polyp.
Withdrawal time among 3 groups. | 6 months
  Withdrawal time from ileocecum, not including the time of treatment and biopsy for polyps.
Caecal intubation rate among 3 groups. | 6 months
  Caecal intubation rate is defined the proportion of patients with caecal intubation.

CONTACTS AND LOCATIONS:
Overall Officials: li yanqing, PhD,MD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China